CLINICAL TRIAL: NCT06070051
Title: A Phase 1b Multi-Center, Open-Label, Dose-Escalation, Prime And Boost Vaccination Evaluation of VRON-0200 Using Two Chimpanzee Adenoviral Vectors in Adult Participants With Chronic HBV Infection Who Are Currently Receiving HBV Nucleos(t)Ide Reverse Transcriptase Inhibitors
Brief Title: Dose-Escalation Prime/Boost Therapeutic Vaccination Study Of 2 Chimp Adenoviral Vectors in Adults With Chronic HBV On Nucleos(t)Ide Therapy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Virion Therapeutics (Industry)
Collaborators: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-0200-101
Record Dates: First submitted 2023-09-20; First posted 2023-10-06 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Chronic Hepatitis B
Keywords: Hep B; Chronic Hep B; HBV; Hepatitis B Virus; Chronic Hepatitis B Virus; CHB; VRON-0200; Virion; therapeutic vaccine; VIR-2218; VIR-3434; Functional cure; Hepatitis B; Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1a: Low Dose VRON-0200-AdC7 Prime, VRON-0200-AdC6 Boost (Experimental): Participants assigned to Cohort 1a will receive a low dose prime vaccination of AdC7 vector on Day 1. They will receive a low dose boost vaccination of vector AdC6 on Day 91.
  Interventions: Biological: VRON-0200-AdC6; Biological: VRON-0200-AdC7
- Cohort 1b: Low Dose VRON-0200-AdC6 Prime, No Boost (Experimental): Participants assigned to Cohort 1b will receive a low dose prime vaccination of AdC6 vector on Day 1. They will not receive a booster vaccination.
  Interventions: Biological: VRON-0200-AdC6
- Cohort 2a: High Dose VRON-0200-AdC7 Prime, VRON-0200-AdC6 Boost (Experimental): Participants assigned to Cohort 2a will receive a high dose prime vaccination of AdC7 vector on Day 1. They will receive a high dose boost vaccination of AdC6 vector on Day 91.
  Interventions: Biological: VRON-0200-AdC6; Biological: VRON-0200-AdC7
- Cohort 2b: High Dose VRON-0200-AdC6 Prime, No Boost (Experimental): Participants assigned to Cohort 2b will receive a high dose prime vaccination of AdC6 vector on Day 1. They will not receive a booster vaccination.
  Interventions: Biological: VRON-0200-AdC6
- Cohort 3a: High Dose VRON-0200-AdC7 Prime, 6 Doses VIR-2218 + VIR-3434, VRON-0200-AdC6 Boost (Experimental): Participants assigned to Cohort 3a will receive a high dose prime vaccination of AdC7 vector on Day 1. They will receive VIR-2218 and VIR-3434 on Days 28, 56, 84, 112, 140, and 168. They will receive a high dose boost vaccination of AdC6 vector on Day 91.
  Interventions: Biological: VRON-0200-AdC6; Biological: VRON-0200-AdC7; Drug: VIR-2218; Drug: VIR-3434
- Cohort 3b: High Dose VRON-0200-AdC7 Prime, 6 Doses VIR-2218 + VIR-3434, No Boost (Experimental): Participants assigned to Cohort 3a will receive a high dose prime vaccination of AdC7 vector on Day 1. They will receive VIR-2218 and VIR-3434 on Days 28, 56, 84, 112, 140, and 168. They will not receive a boost vaccination.
  Interventions: Biological: VRON-0200-AdC7; Drug: VIR-2218; Drug: VIR-3434

INTERVENTIONS:
Biological: VRON-0200-AdC6 — VRON-0200 chimpanzee adenovirus serotype 6 vaccine vector
  Arms: Cohort 1a: Low Dose VRON-0200-AdC7 Prime, VRON-0200-AdC6 Boost; Cohort 1b: Low Dose VRON-0200-AdC6 Prime, No Boost; Cohort 2a: High Dose VRON-0200-AdC7 Prime, VRON-0200-AdC6 Boost; Cohort 2b: High Dose VRON-0200-AdC6 Prime, No Boost; Cohort 3a: High Dose VRON-0200-AdC7 Prime, 6 Doses VIR-2218 + VIR-3434, VRON-0200-AdC6 Boost
Biological: VRON-0200-AdC7 — VRON-0200 chimpanzee adenovirus serotype 7 vaccine vector
  Arms: Cohort 1a: Low Dose VRON-0200-AdC7 Prime, VRON-0200-AdC6 Boost; Cohort 2a: High Dose VRON-0200-AdC7 Prime, VRON-0200-AdC6 Boost; Cohort 3a: High Dose VRON-0200-AdC7 Prime, 6 Doses VIR-2218 + VIR-3434, VRON-0200-AdC6 Boost; Cohort 3b: High Dose VRON-0200-AdC7 Prime, 6 Doses VIR-2218 + VIR-3434, No Boost
Drug: VIR-2218 — VIR-2218 given by subcutaneous injection
  Other Names: elebsiran
  Arms: Cohort 3a: High Dose VRON-0200-AdC7 Prime, 6 Doses VIR-2218 + VIR-3434, VRON-0200-AdC6 Boost; Cohort 3b: High Dose VRON-0200-AdC7 Prime, 6 Doses VIR-2218 + VIR-3434, No Boost
Drug: VIR-3434 — VIR-3434 given by subcutaneous injection
  Other Names: tobevibart; BRII-877
  Arms: Cohort 3a: High Dose VRON-0200-AdC7 Prime, 6 Doses VIR-2218 + VIR-3434, VRON-0200-AdC6 Boost; Cohort 3b: High Dose VRON-0200-AdC7 Prime, 6 Doses VIR-2218 + VIR-3434, No Boost

SUMMARY:
This Phase 1b clinical study is a multi-center, open-label, dose escalation, prime only, and prime plus boost therapeutic vaccination study of 2 distinct chimpanzee adenoviral vectors (AdC6 and AdC7), containing parts of hepatitis B virus (HBV) core and polymerase antigens fused within glycoprotein D in a cohort of chronic hepatitis B (CHB)-infected adult participants who are currently receiving entecavir, tenofovir (tenofovir alafenamide fumarate or tenofovir disoproxil fumarate), or lamivudine, with documented HBV viral load suppression for at least 12 months.

Approximately 24 participants will be enrolled in Group 1 and randomized to Cohort 1a or Cohort 1b. Those assigned to Cohort 1a will receive a low dose prime therapeutic vaccination of vector AdC7 on Day 1, followed by a booster vaccination on Day 91 using vector AdC6. Those assigned to Cohort 1b will receive a low dose prime therapeutic vaccination of vector AdC6 on Day 1, and will not receive a booster vaccination.

Group 2 will then enroll approximately 24 participants randomized to Cohort 2a or Cohort 2b. Those assigned to Cohort 2a will receive a high dose prime therapeutic vaccination of vector AdC7 on Day 1, followed by a booster vaccination on Day 91 using vector AdC6. Those assigned to Cohort 2b will receive a high dose prime therapeutic vaccination of vector AdC6 on Day 1, and will not receive a booster vaccination.

Group 3 will enroll approximately 8 participants randomized into Cohort 3a or Cohort 3b. Cohort 3a will receive the high dose prime VRON-0200 vaccination of vector AdC7 on Day 1, followed by doses of VIR-2218 plus VIR-3434 on Days 28, 56, 84, 112, 140 and 168, and then a booster using a high dose VRON-0200 vaccination of vector AdC6 on Day 196. Cohort 3b will receive the same high dose prime VRON-0200 vaccination of vector AdC7 followed by 6 doses of VIR-2218 plus VIR-3434 at the same timepoints as Cohort 3a, but will not receive the booster dose on Day 196.

VRON-0200 vaccine doses will be administered by intramuscular (IM) injection. VIR-2218 and VIR-3434 will be administered subcutaneously.

All study participants will be followed for a total of 1 year post-prime vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Documented chronic HBV infection (eg, HBsAg+ ≥ 6 months with detectable HBsAg at screening)
2. Receipt of either entecavir, tenofovir (tenofovir alafenamide fumarate or tenofovir disoproxil fumarate), or lamivudine for at least 12 months before screening with no reported antiviral resistance during this time; still on treatment at screening and expected to stay on therapy during the study period
3. Virally suppressed for > 12 months (HBV DNA < 40 IU/mL)
4. No clinical diagnosis of advanced liver fibrosis and/or cirrhosis

Exclusion Criteria:

1. History of hepatic decompensation, advanced fibrosis, or liver transplantation
2. History of hepatocellular carcinoma
3. History of risk factors for thrombosis and thrombocytopenia
4. Documented hepatitis A, hepatitis C, hepatitis D, hepatitis E, or HIV (or history of prior active disease)
5. Pregnant, nursing, or planning a pregnancy during the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events | 28 days
  Number and percent of participants with 1 or more treatment-emergent adverse events within 28 days after the last dose by cohort.
Grade 3 Adverse Events | 28 days
  Number and percent of participants with Grade 3 or higher local and/or systemic reactions within 28 days after the last dose by cohort.
Clinically Significant Changes in Lab Values | 28 days
  Number and percent of participants with clinically significant changes from pre-vaccination laboratory values within 28 days after the last dose by cohort.
Serious Adverse Events | 6 months
  Number and percent of participants with serious adverse events within 6 months after the last dose by cohort.
Medically Attended Adverse Events | 6 months
  Number and percent of participants with medically attended adverse events within 6 months after the last dose by cohort.

SECONDARY OUTCOMES:
Adverse Events | 360 days
  Number and percentage of adverse events for all participants through Day 360.
T Cell Frequencies | 360 days
  Change from baseline in vaccine-induced CD8+ T cell frequencies in the blood.

OTHER OUTCOMES:
Hepatitis B Virus DNA | 360 days
  Quantitative changes from baseline over time in HBV DNA
Hepatitis B Virus Pregenomic RNA | 360 days
  Quantitative changes from baseline over time in HBV pgRNA
Hepatitis B Surface Antigen | 360 days
  Quantitative changes from baseline over time in HBsAg

CONTACTS AND LOCATIONS:
Overall Officials: Sue Currie, PhD, Study Director — Virion Therapeutics
Locations (3):
- Chinese University of Hong Kong, Hong Kong, Hong Kong
- New Zealand (2):
  - Aotearoa Clinical Trials, Middlemore Hospital, Auckland
  - Auckland City Hospital, Auckland